CLINICAL TRIAL: NCT00338884
Title: A Phase II Efficacy And Safety Study Of Sunitinib Malate (SU011248) Administered In A Continuous Daily Regimen In Patients With Advanced (First-Line) Renal Cell Cancer
Brief Title: Safety And Effectiveness Of Daily Dosing With 37.5 mg Sunitinib Malate In Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181110
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

ARMS (1):
- SUNITINIB MALATE. (Experimental): Sunitinib malate starting dose 37.5 mg daily continuous daily schedule
  Interventions: Drug: Sunitinib malate

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib malate starting dose 37.5 mg daily continuous daily schedule

SUMMARY:
A phase II study to allow patients with advanced kidney cancer access to sunitinib malate treatment and to find out the good and bad effects of taking 37.5 mg sunitinib malate in a continuous daily regimen (once per day) for one year.

ELIGIBILITY:
Inclusion Criteria:

* Advanced kidney cancer

Exclusion Criteria:

* Previous treatment for kidney cancer, except surgical removal of kidney tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Argentina (3):
  - Pfizer Investigational Site, Córdoba, Córdoba Province
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
- Australia (3):
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, East Bentleigh, Victoria
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Mexico (2):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (3):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei

REFERENCES:
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Grunwald V, McKay RR, Krajewski KM, Kalanovic D, Lin X, Perkins JJ, Simantov R, Choueiri TK. Depth of remission is a prognostic factor for survival in patients with metastatic renal cell carcinoma. Eur Urol. 2015 May;67(5):952-8. doi: 10.1016/j.eururo.2014.12.036. Epub 2015 Jan 7. PMID 25577718
- [Derived] Barrios CH, Hernandez-Barajas D, Brown MP, Lee SH, Fein L, Liu JH, Hariharan S, Martell BA, Yuan J, Bello A, Wang Z, Mundayat R, Rha SY. Phase II trial of continuous once-daily dosing of sunitinib as first-line treatment in patients with metastatic renal cell carcinoma. Cancer. 2012 Mar 1;118(5):1252-9. doi: 10.1002/cncr.26440. Epub 2011 Sep 6. PMID 21898376
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181110&StudyName=Safety%20And%20Effectiveness%20Of%20Daily%20Dosing%20With%2037.5%20mg%20Sunitinib%20Malate%20In%20Patients%20With%20Advanced%20Kidney%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: 37.5 milligrams (mg) oral sunitinib malate. Dose could have been reduced to 25 mg daily due to sunitinib related toxicities.
Period: Overall Study
Arm/Group | Sunitinib
Started | 120
Received Treatment | 119
Completed | 42
Not Completed | 78
Not completed — Objective Disease Progression or Relapse | 44
Not completed — Adverse Event | 14
Not completed — Death | 8
Not completed — Other | 4
Not completed — Global Deterioration of Health Status | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Randomized But Did Not Receive Treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib: 37.5 mg oral sunitinib malate. Dose could have been reduced to 25 mg daily due to sunitinib related toxicities.
Arm/Group | Sunitinib
Number analyzed (Participants) | 119
Age, Customized [Number; unit: participants]
  18 to 44 years | 14
  45 to 64 years | 69
  > = 65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Overall Confirmed Objective Response (OR)
Description: OR = subjects with confirmed complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) persisting > = 4 weeks after initial documentation of response. A CR was defined as the disappearance of all target lesions. A PR was defined as a ≥ 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From start of treatment through Day 1 of Weeks 5, 9, and every 8 weeks thereafter
Population: Safety Population=all enrolled subjects who received at least 1 dose of sunitinib. For OR rate analysis, subjects who did not have a baseline assessment of disease were excluded from the analysis. Number of participants analyzed = number of subjects evaluable for OR analysis.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 116
participants | 41
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 35.3, 95% CI 2-sided [26.7 to 44.8] — ORR=proportion of subjects with confirmed CR or PR, relative to total subjects who received at least 1 dose of study medication, had a baseline disease assessment, and had the correct histological cancer type

2. Secondary Outcome: Duration of Response (DR)
Description: Time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death due to to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. DR was calculated as [the end date for DR minus first CR or PR that was subsequently confirmed +1]/7.
Time Frame: From start of treatment through Day 1 of Weeks 5, 9, and every 8 weeks thereafter or death due to any cause
Population: Safety population subgroup of subjects with a confirmed objective tumor response. DR was only calculated for the subgroup of subjects with a confirmed objective response.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 41
months | 7.14 [6.28 to 8.00]

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time from date of first dose of study medication to first documentation of objective tumor progression. The 50% quartile point estimate is provided. The criteria for tumor progression was according to RECIST.
Time Frame: From start of treatment through Day 1 of Weeks 5, 9, and every 8 weeks thereafter
Population: Safety population. 64 subjects were censored. Number of participants analyzed = number of subjects evaluable for tumor progression analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 118
months | 10.0 [7.2 to NA] — The upper confidence interval was not reached.

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from start of study medication to first documentation of objective tumor progression or to death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. PFS (in months) was calculated as (first event date minus first dose date +1)/7.
Time Frame: From start of treatment through Day 1 of Weeks 5, 9, and every 8 weeks thereafter or death
Population: Safety population. Number of participants analyzed = number of subjects evaluable for PFS analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 118
months | 9.0 [5.6 to 11.1]

5. Secondary Outcome: 1-Year Survival
Description: One year survival rate defined as the probability that a subject was alive 1 year after the date of first study treatment.
Time Frame: From start of treatment through Day 1 of Weeks 5, 9, and every 8 weeks thereafter up until 1 year
Population: Safety population. Number of participants analyzed = number of subjects evaluable for 1 year survival analysis.
Measure: Median (95% Confidence Interval); unit: percent chance of survival
Arm/Group | Sunitinib
Number analyzed (Participants) | 118
percent chance of survival | 67.8 [59.2 to 76.3]

6. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of Sunitinib
Description: Ctrough = the concentration prior to study drug administration.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: Pharmacokinetic (PK) population = treated and had least 1 PK sample taken. Number of Participants analyzed = number of subjects evaluable for PK analysis. n=number of subjects evaluable at each time point.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Sunitinib
Number analyzed (Participants) | 111
nanograms (ng)/milliliter (mL)
  Day 1, Week 1 (n=111) | 7.15 (18.80)
  Day 1, Week 3 (n=108) | 54.78 (23.67)
  Day 1, Week 5 (n=106) | 45.64 (22.83)
  Day 1, Week 7 (n=104) | 46.35 (21.98)
  Day 1, Week 9 (n=97) | 47.54 (24.96)
  Day 1, Week 13 (n=93) | 41.29 (22.41)
  Day 1, Week 17 (n=82) | 41.65 (20.25)
  Day 1, Week 21 (n=73) | 35.95 (20.38)
  Day 1, Week 25 (n=70) | 36.39 (20.72)
  Day 1, Week 29 (n=58) | 38.01 (21.24)
  Day 1, Week 33 (n=58) | 33.72 (18.94)
  Day 1, Week 37 (n=50) | 36.04 (16.48)
  Day 1, Week 41 (n=49) | 33.33 (15.80)
  Day 1, Week 45 (n=44) | 36.20 (13.79)
  Day 1, Week 49 (n=40) | 36.49 (13.10)
  Day 1, Week 53 (n=33) | 33.10 (16.18)

7. Secondary Outcome: Ctrough Stratified by CR or PR Versus Progressive Disease (PD) for Sunitinib
Description: Summary statistics of ctrough at each time point by group (CR or PR versus PD) are presented.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: PK. Number of Participants analyzed = number of subjects with evaluable PK data and tumor response at baseline. n=number of subjects with evaluable PK data and tumor response at each specified time point. No subjects had PD following Week 33.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 41
ng/mL
  Day 1, Week 1 (CR or PR, n=39) | 0.000 [0 to 71.3]
  Day 1, Week 3 (CR or PR, n=40) | 57.900 [16.9 to 109]
  Day 1, Week 5 (CR or PR, n=38) | 45.000 [2.02 to 93.6]
  Day 1, Week 7 (CR or PR, n=40) | 45.400 [18.5 to 83.9]
  Day 1, Week 9 (CR or PR, n=38) | 46.250 [0 to 74]
  Day 1, Week 13 (CR or PR, n=41) | 40.000 [2.13 to 91.4]
  Day 1, Week 17 (CR or PR, n=38) | 41.350 [0 to 83]
  Day 1, Week 21 (CR or PR, n=38) | 34.400 [0 to 99.7]
  Day 1, Week 25 (CR or PR, n=37) | 34.200 [0 to 92.7]
  Day 1, Week 29 (CR or PR, n=32) | 34.450 [5.91 to 128]
  Day 1, Week 33 (CR or PR, n=33) | 33.000 [0 to 64.9]
  Day 1, Week 37 (CR or PR, n=28) | 35.350 [4.1 to 73.3]
  Day 1, Week 41 (CR or PR, n=28) | 30.900 [6.15 to 77]
  Day 1, Week 45 (CR or PR, n=29) | 34.000 [6.87 to 64.9]
  Day 1, Week 49 (CR or PR, n=26) | 36.250 [6.97 to 69.7]
  Day 1, Week 53 (CR or PR, n=21) | 28.600 [0 to 72.6]
  Day 1, Week 1 (PD, n=16) | 0.000 [0 to 51.1]
  Day 1, Week 3 (PD, n=15) | 50.200 [0 to 150]
  Day 1, Week 5 (PD, n=15) | 45.600 [6.81 to 88.7]
  Day 1, Week 7 (PD, n=13) | 35.600 [0 to 69.5]
  Day 1, Week 9 (PD, n=8) | 39.050 [0 to 70.7]
  Day 1, Week 13 (PD, n=1) | 25.100 [25.1 to 25.1]
  Day 1, Week 17 (PD, n=1) | 28.200 [28.2 to 28.2]
  Day 1, Week 21 (PD, n=1) | 47.700 [47.7 to 47.7]
  Day 1, Week 25 (PD, n=1) | 22.700 [22.7 to 22.7]
  Day 1, Week 29 (PD, n=1) | 23.700 [23.7 to 23.7]
  Day 1, Week 33 (PD, n=1) | 9.520 [9.52 to 9.52]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 1 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5581, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 3 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.7635, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 5 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8366, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 7 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.0278, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 9 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.1988, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 13 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2898, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 17 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3567, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 21 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4547, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 25 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2809, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 29 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3259, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Sunitinib; Day 1, Week 33 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2702, Wilcoxon Rank Sum Test

8. Secondary Outcome: Ctrough Stratified by Tumor Response (CR or PR or [Stable Disease (SD) > = 12 Weeks] Versus PD) for Sunitinib
Description: Summary statistics of ctrough at each time point by group (CR or PR or SD versus PD) are presented.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: as for outcome 7
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 88
ng/mL
  Day 1, Week 1 (CR or PR or SD, n=83) | 0.000 [0 to 88.4]
  Day 1, Week 3 (CR or PR or SD, n=83) | 55.300 [16.9 to 114]
  Day 1, Week 5 (CR or PR or SD, n=83) | 44.600 [1.39 to 96.8]
  Day 1, Week 7 (CR or PR or SD, n=86) | 46.750 [0 to 118]
  Day 1, Week 9 (CR or PR or SD, n=85) | 49.500 [0 to 150]
  Day 1, Week 13 (CR or PR or SD, n=88) | 39.550 [0 to 106]
  Day 1, Week 17 (CR or PR or SD, n=79) | 42.300 [0 to 132]
  Day 1, Week 21 (CR or PR or SD, n=71) | 36.500 [0 to 99.7]
  Day 1, Week 25 (CR or PR or SD, n=68) | 35.500 [0 to 92.7]
  Day 1, Week 29 (CR or PR or SD, n=56) | 37.250 [0 to 128]
  Day 1, Week 33 (CR or PR or SD, n=56) | 34.400 [0 to 102]
  Day 1, Week 37 (CR or PR or SD, n=49) | 35.300 [4.1 to 74.2]
  Day 1, Week 41 (CR or PR or SD, n=49) | 33.200 [0 to 77]
  Day 1, Week 45 (CR or PR or SD, n=44) | 35.950 [1.96 to 64.9]
  Day 1, Week 49 (CR or PR or SD, n=40) | 37.250 [6.97 to 69.7]
  Day 1, Week 53 (CR or PR or SD, n=32) | 31.100 [0 to 72.6]
  Day 1, Week 1 (PD, n=16) | 0.000 [0 to 51.1]
  Day 1, Week 3 (PD, n=15) | 50.200 [0 to 150]
  Day 1, Week 5 (PD, n=15) | 45.600 [6.81 to 88.7]
  Day 1, Week 7 (PD, n=13) | 35.600 [0 to 69.5]
  Day 1, Week 9 (PD, n=8) | 39.050 [0 to 70.7]
  Day 1, Week 13 (PD, n=1) | 25.100 [25.1 to 25.1]
  Day 1, Week 17 (PD, n=1) | 28.200 [28.2 to 28.2]
  Day 1, Week 21 (PD, n=1) | 47.700 [47.7 to 47.7]
  Day 1, Week 25 (PD, n=1) | 22.700 [22.7 to 22.7]
  Day 1, Week 29 (PD, n=1) | 23.700 [23.7 to 23.7]
  Day 1, Week 33 (PD, n=1) | 9.520 [9.52 to 9.52]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 1 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.7154, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 3 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.6263, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 5 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.9608, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 7 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.0300, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 9 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.0927, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 13 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2873, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 17 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3018, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 21 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.4161, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 25 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3069, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 29 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2920, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Sunitinib; Day 1, Week 33 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2409, Wilcoxon Rank Sum Test

9. Secondary Outcome: Ctrough of SU-012662 (Sunitinib's Metabolite)
Description: Ctrough = the concentration prior to study drug administration.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: PK. Number of Participants analyzed = number of subjects evaluable for PK analysis. n=number of subjects evaluable at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 111
ng/mL
  Day 1, Week 1 (n=111) | 2.62 (6.88)
  Day 1, Week 3 (n=108) | 20.27 (8.17)
  Day 1, Week 5 (n=106) | 20.25 (11.73)
  Day 1, Week 7 (n=104) | 20.41 (12.45)
  Day 1, Week 9 (n=97) | 21.18 (13.07)
  Day 1, Week 13 (n=93) | 20.01 (13.88)
  Day 1, Week 17 (n=82) | 19.76 (12.84)
  Day 1, Week 21 (n=73) | 17.13 (11.64)
  Day 1, Week 25 (n=70) | 17.30 (12.75)
  Day 1, Week 29 (n=58) | 17.38 (11.76)
  Day 1, Week 33 (n=58) | 16.55 (12.20)
  Day 1, Week 37 (n=50) | 15.71 (6.70)
  Day 1, Week 41 (n=49) | 16.50 (8.95)
  Day 1, Week 45 (n=44) | 15.61 (7.66)
  Day 1, Week 49 (n=40) | 16.57 (7.65)
  Day 1, Week 53 (n=33) | 13.81 (7.21)

10. Secondary Outcome: Ctrough Stratified by CR or PR Versus PD for SU-012662 (Sunitinib's Metabolite)
Description: Summary statistics of ctrough at each time point by group (CR or PR versus PD) are presented.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: as for outcome 7
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 41
ng/mL
  Day 1, Week 1 (CR or PR, n=39) | 0.000 [0 to 23.8]
  Day 1, Week 3 (CR or PR, n=40) | 18.250 [6.75 to 36.1]
  Day 1, Week 5 (CR or PR, n=38) | 16.650 [2.34 to 41.2]
  Day 1, Week 7 (CR or PR, n=40) | 17.300 [7.18 to 46.6]
  Day 1, Week 9 (CR or PR, n=38) | 15.100 [0 to 45.2]
  Day 1, Week 13 (CR or PR, n=41) | 15.900 [3.54 to 81.9]
  Day 1, Week 17 (CR or PR, n=38) | 14.300 [0 to 45.3]
  Day 1, Week 21 (CR or PR, n=38) | 12.600 [0 to 52.1]
  Day 1, Week 25 (CR or PR, n=37) | 14.500 [0 to 80.3]
  Day 1, Week 29 (CR or PR, n=32) | 12.850 [3.23 to 60.3]
  Day 1, Week 33 (CR or PR, n=33) | 12.800 [1.01 to 31.4]
  Day 1, Week 37 (CR or PR, n=28) | 14.350 [4.52 to 31]
  Day 1, Week 41 (CR or PR, n=28) | 14.000 [6.31 to 40.8]
  Day 1, Week 45 (CR or PR, n=29) | 13.400 [6.08 to 39.2]
  Day 1, Week 49 (CR or PR, n=26) | 14.700 [4.62 to 33.1]
  Day 1, Week 53 (CR or PR, n=21) | 11.600 [0 to 24.6]
  Day 1, Week 1 (PD, n=16) | 0.000 [0 to 16.6]
  Day 1, Week 3 (PD, n=15) | 20.000 [0 to 39.7]
  Day 1, Week 5 (PD, n=15) | 18.800 [5.81 to 49.1]
  Day 1, Week 7 (PD, n=13) | 14.300 [0 to 58.5]
  Day 1, Week 9 (PD, n=8) | 16.550 [0 to 54.1]
  Day 1, Week 13 (PD, n=1) | 9.710 [9.71 to 9.71]
  Day 1, Week 17 (PD, n=1) | 12.600 [12.6 to 12.6]
  Day 1, Week 21 (PD, n=1) | 23.400 [23.4 to 23.4]
  Day 1, Week 25 (PD, n=1) | 29.400 [29.4 to 29.4]
  Day 1, Week 29 (PD, n=1) | 13.700 [13.7 to 13.7]
  Day 1, Week 33 (PD, n=1) | 4.360 [4.36 to 4.36]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 1 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5784, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 3 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.6251, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 5 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.1639, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 7 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2782, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 9 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8627, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 13 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4620, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 17 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.7575, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 21 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3566, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 25 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2809, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 29 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8758, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Sunitinib; Day 1, Week 33 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2702, Wilcoxon Rank Sum Test

11. Secondary Outcome: Ctrough Stratified by Tumor Response (CR or PR or [SD > = 12 Weeks] Versus PD) for SU-012662 (Sunitinib's Metabolite)
Description: Summary statistics of ctrough at each time point by group (CR or PR or SD versus PD) are presented.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: as for outcome 7
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 88
ng/mL
  Day 1, Week 1 (CR or PR or SD, n=83) | 0.000 [0 to 34.6]
  Day 1, Week 3 (CR or PR or SD, n=83) | 18.800 [6.75 to 54.1]
  Day 1, Week 5 (CR or PR or SD, n=83) | 17.300 [0 to 70.6]
  Day 1, Week 7 (CR or PR or SD, n=86) | 17.900 [0 to 76.3]
  Day 1, Week 9 (CR or PR or SD, n=85) | 18.700 [0 to 57.7]
  Day 1, Week 13 (CR or PR or SD, n=88) | 16.350 [1.31 to 81.9]
  Day 1, Week 17 (CR or PR or SD, n=79) | 14.600 [0 to 61.1]
  Day 1, Week 21 (CR or PR or SD, n=71) | 14.100 [0 to 52.8]
  Day 1, Week 25 (CR or PR or SD, n=68) | 14.950 [0 to 80.3]
  Day 1, Week 29 (CR or PR or SD, n=56) | 14.900 [0 to 60.3]
  Day 1, Week 33 (CR or PR or SD, n=56) | 14.050 [1.01 to 71.9]
  Day 1, Week 37 (CR or PR or SD, n=49) | 15.500 [4.52 to 36.2]
  Day 1, Week 41 (CR or PR or SD, n=49) | 15.400 [0 to 43.5]
  Day 1, Week 45 (CR or PR or SD, n=44) | 13.700 [6.08 to 39.2]
  Day 1, Week 49 (CR or PR or SD, n=40) | 14.700 [4.62 to 42.9]
  Day 1, Week 53 (CR or PR or SD, n=32) | 11.450 [0 to 27.1]
  Day 1, Week 1 (PD, n=16) | 0.000 [0 to 16.6]
  Day 1, Week 3 (PD, n=15) | 20.000 [0 to 39.7]
  Day 1, Week 5 (PD, n=15) | 18.800 [5.81 to 49.1]
  Day 1, Week 7 (PD, n=13) | 14.300 [0 to 58.5]
  Day 1, Week 9 (PD, n=8) | 16.550 [0 to 54.1]
  Day 1, Week 13 (PD, n=1) | 9.710 [9.71 to 9.71]
  Day 1, Week 17 (PD, n=1) | 12.600 [12.6 to 12.6]
  Day 1, Week 21 (PD, n=1) | 23.400 [23.4 to 23.4]
  Day 1, Week 25 (PD, n=1) | 29.400 [29.4 to 29.4]
  Day 1, Week 29 (PD, n=1) | 13.700 [13.7 to 13.7]
  Day 1, Week 33 (PD, n=1) | 4.360 [4.36 to 4.36]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 1 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.7267, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 3 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.8555, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 5 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2259, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 7 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2074, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 9 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.4779, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 13 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3628, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 17 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.5460, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 21 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3637, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 25 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2229, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 29 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.9759, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Sunitinib; Day 1, Week 33 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2179, Wilcoxon Rank Sum Test

12. Secondary Outcome: Ctrough of Total Drug (Sunitinib + SU-012662)
Description: Ctrough = the concentration prior to study drug administration.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 111
ng/mL
  Day 1, Week 1 (n=111) | 9.77 (25.09)
  Day 1, Week 3 (n=108) | 75.04 (29.48)
  Day 1, Week 5 (n=106) | 65.89 (32.37)
  Day 1, Week 7 (n=104) | 66.76 (32.03)
  Day 1, Week 9 (n=97) | 68.72 (35.01)
  Day 1, Week 13 (n=93) | 61.31 (33.31)
  Day 1, Week 17 (n=82) | 61.41 (30.43)
  Day 1, Week 21 (n=73) | 53.09 (30.50)
  Day 1, Week 25 (n=70) | 53.69 (31.52)
  Day 1, Week 29 (n=58) | 55.39 (31.40)
  Day 1, Week 33 (n=58) | 50.27 (29.55)
  Day 1, Week 37 (n=50) | 51.74 (20.54)
  Day 1, Week 41 (n=49) | 49.83 (23.68)
  Day 1, Week 45 (n=44) | 51.82 (19.15)
  Day 1, Week 49 (n=40) | 53.07 (18.25)
  Day 1, Week 53 (n=33) | 46.91 (21.56)

13. Secondary Outcome: Ctrough Stratified by CR or PR Versus PD for Total Drug (Sunitinib + SU012662)
Description: Summary statistics of ctrough at each time point by group (CR or PR versus PD) are presented.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: as for outcome 7
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 41
ng/mL
  Day 1, Week 1 (CR or PR, n=39) | 0.000 [0 to 95.1]
  Day 1, Week 3 (CR or PR, n=40) | 76.950 [23.65 to 139.9]
  Day 1, Week 5 (CR or PR, n=38) | 65.900 [4.36 to 125.5]
  Day 1, Week 7 (CR or PR, n=40) | 66.100 [28.02 to 120.4]
  Day 1, Week 9 (CR or PR, n=38) | 65.150 [0 to 118.3]
  Day 1, Week 13 (CR or PR, n=41) | 57.600 [5.67 to 158.5]
  Day 1, Week 17 (CR or PR, n=38) | 55.660 [0 to 128.2]
  Day 1, Week 21 (CR or PR, n=38) | 47.370 [0 to 135.3]
  Day 1, Week 25 (CR or PR, n=37) | 50.700 [0 to 173]
  Day 1, Week 29 (CR or PR, n=32) | 50.650 [10.78 to 185]
  Day 1, Week 33 (CR or PR, n=33) | 46.000 [1.01 to 85.5]
  Day 1, Week 37 (CR or PR, n=28) | 49.750 [8.62 to 98.9]
  Day 1, Week 41 (CR or PR, n=28) | 43.365 [12.46 to 106]
  Day 1, Week 45 (CR or PR, n=29) | 45.200 [14.39 to 102.6]
  Day 1, Week 49 (CR or PR, n=26) | 49.975 [11.59 to 89]
  Day 1, Week 53 (CR or PR, n=21) | 41.000 [0 to 90.5]
  Day 1, Week 1 (PD, n=16) | 0.000 [0 to 67.7]
  Day 1, Week 3 (PD, n=15) | 69.000 [0 to 183]
  Day 1, Week 5 (PD, n=15) | 64.700 [12.62 to 129.6]
  Day 1, Week 7 (PD, n=13) | 50.200 [0 to 128]
  Day 1, Week 9 (PD, n=8) | 55.850 [0 to 124.8]
  Day 1, Week 13 (PD, n=1) | 34.810 [34.81 to 34.81]
  Day 1, Week 17 (PD, n=1) | 40.800 [40.8 to 40.8]
  Day 1, Week 21 (PD, n=1) | 71.100 [71.1 to 71.1]
  Day 1, Week 25 (PD, n=1) | 52.100 [52.1 to 52.1]
  Day 1, Week 29 (PD, n=1) | 37.400 [37.4 to 37.4]
  Day 1, Week 33 (PD, n=1) | 13.880 [13.88 to 13.88]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 1 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5784, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 3 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.9625, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 5 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8519, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 7 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.0513, Wilcoxon Rank Sum Test; Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 9 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4051, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 13 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2548, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 17 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5091, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 21 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3133, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 25 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.9278, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 29 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4070, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Sunitinib; Day 1, Week 33 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.2703, Wilcoxon Rank Sum Test

14. Secondary Outcome: Ctrough Stratified by Tumor Response (CR or PR or [SD > = 12 Weeks] Versus PD) for Total Drug (Sunitinib + SU012662)
Description: Summary statistics of ctrough at each time point by group (CR or PR or SD versus PD) are presented.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: as for outcome 7
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 88
ng/mL
  Day 1, Week 1 (CR or PR or SD, n=83) | 0.000 [0 to 103.3]
  Day 1, Week 3 (CR or PR or SD, n=83) | 75.000 [23.65 to 166.1]
  Day 1, Week 5 (CR or PR or SD, n=83) | 63.300 [1.47 to 157.6]
  Day 1, Week 7 (CR or PR or SD, n=86) | 66.400 [0 to 194.3]
  Day 1, Week 9 (CR or PR or SD, n=85) | 70.600 [0 to 201.4]
  Day 1, Week 13 (CR or PR or SD, n=88) | 57.600 [1.31 to 158.5]
  Day 1, Week 17 (CR or PR or SD, n=79) | 58.100 [0 to 183.5]
  Day 1, Week 21 (CR or PR or SD, n=71) | 49.860 [0 to 135.3]
  Day 1, Week 25 (CR or PR or SD, n=68) | 51.150 [0 to 173]
  Day 1, Week 29 (CR or PR or SD, n=56) | 53.500 [0 to 185]
  Day 1, Week 33 (CR or PR or SD, n=56) | 50.050 [1.01 to 173.9]
  Day 1, Week 37 (CR or PR or SD, n=49) | 50.800 [8.62 to 102.4]
  Day 1, Week 41 (CR or PR or SD, n=49) | 48.000 [0 to 106]
  Day 1, Week 45 (CR or PR or SD, n=44) | 50.500 [9.93 to 102.6]
  Day 1, Week 49 (CR or PR or SD, n=40) | 54.885 [11.59 to 89]
  Day 1, Week 53 (CR or PR or SD, n=32) | 42.160 [0 to 90.5]
  Day 1, Week 1 (PD, n=16) | 0.000 [0 to 67.7]
  Day 1, Week 3 (PD, n=15) | 69.000 [0 to 183]
  Day 1, Week 5 (PD, n=15) | 64.700 [12.62 to 129.6]
  Day 1, Week 7 (PD, n=13) | 50.200 [0 to 128]
  Day 1, Week 9 (PD, n=8) | 55.850 [0 to 124.8]
  Day 1, Week 13 (PD, n=1) | 34.810 [34.81 to 34.81]
  Day 1, Week 17 (PD, n=1) | 40.800 [40.8 to 40.8]
  Day 1, Week 21 (PD, n=1) | 71.100 [71.1 to 71.1]
  Day 1, Week 25 (PD, n=1) | 52.100 [52.1 to 52.1]
  Day 1, Week 29 (PD, n=1) | 37.400 [37.4 to 37.4]
  Day 1, Week 33 (PD, n=1) | 13.880 [13.88 to 13.88]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 1 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.7267, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 3 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.8286, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 5 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.6867, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 7 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.0450, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 9 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.1740, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 13 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2703, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 17 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3659, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 21 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3391, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 25 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.9800, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 29 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3350, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: Sunitinib; Day 1, Week 33 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2179, Wilcoxon Rank Sum Test

15. Secondary Outcome: Ctrough Correlated With Serious Adverse Events (SAEs)
Description: Serious adverse event defined as any untoward medical occurrence at any dose that: Results in death; Is life-threatening (immediate risk of death); Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Results in congenital anomaly/birth defect.
Time Frame: Predose on Day 1 of Weeks 1, 3, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, and 53
Population: Ctrough correlation analyses with SAEs were not performed due to low frequency of individual SAEs.
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

16. Secondary Outcome: Vascular Endothelial Growth Factor (VEGF) Concentration at Baseline
Time Frame: Baseline
Population: Safety population. Number of Participants analyzed = number of subjects with evaluable data at baseline.
Measure: Mean (Standard Deviation); unit: picograms (pg)/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 113
picograms (pg)/mL | 154.8 (186.6)

17. Secondary Outcome: VEGF at Baseline Stratified by Tumor Response (CR or PR Versus PD)
Description: Summary statistics of VEGF at baseline by group (CR or PR versus PD) are presented.
Time Frame: Baseline (Cycle 1, Day 1)
Population: Safety population. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 45
pg/mL
  Cycle 1, Day 1 (CR or PR, n=39) | 73.600 [19.2 to 454.9]
  Cycle 1, Day 1 (PD, n=16) | 109.300 [44.4 to 1199.3]
Statistical Analysis 1: Comparison: Sunitinib; CR or PR Versus PD; Test type: Superiority or Other; p = 0.0680, Wilcoxon Rank Sum Test

18. Secondary Outcome: VEGF at Baseline Stratified by Tumor Response (CR or PR or [SD > = 12 Weeks] Versus PD)
Description: Summary statistics of VEGF at baseline by group (CR or PR or SD versus PD) are presented.
Time Frame: Baseline (Cycle 1, Day 1)
Population: Safety population. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 101
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=85) | 86.400 [14.1 to 624.5]
  Cycle 1, Day 1 (PD, n=16) | 109.300 [44.4 to 1199.3]
Statistical Analysis 1: Comparison: Sunitinib; CR or PR or (SD > = 12 Weeks) Versus PD; Test type: Superiority or Other; p = 0.1159, Wilcoxon Rank Sum Test

19. Secondary Outcome: VEGF Ratio to Baseline at Each Time Point
Description: VEGF concentration at each time point divided by VEGF concentration at baseline (ratio to baseline).
Time Frame: Baseline to Day 1 of Weeks 3 through 53
Population: Safety population. Number of Participants analyzed = number of subjects with evaluable data at baseline. n=number of subjects with evaluable data at each specified time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 113
ratio
  Day 1, Week 3 (n=108) | 2.9 (2.8)
  Day 1, Week 5 (n=104) | 2.6 (2.9)
  Day 1, Week 7 (n=101) | 2.6 (2)
  Day 1, Week 9 (n=95) | 3.4 (3.3)
  Day 1, Week 13 (n=91) | 3.2 (3.4)
  Day 1, Week 17 (n=78) | 2.8 (2.4)
  Day 1, Week 21 (n=70) | 2.6 (2.1)
  Day 1, Week 25 (n=67) | 3 (3.2)
  Day 1, Week 29 (n=55) | 2.5 (1.8)
  Day 1, Week 33 (n=54) | 2.3 (1.4)
  Day 1, Week 37 (n=49) | 2.7 (2.1)
  Day 1, Week 41 (n=48) | 5.5 (20.5)
  Day 1, Week 45 (n=41) | 2.9 (2.1)
  Day 1, Week 49 (n=37) | 2.8 (1.8)
  Day 1, Week 53 (n=30) | 3.2 (3)

20. Secondary Outcome: VEGF Ratio to Baseline Stratified by Tumor Response (CR or PR Versus PD)
Description: Median VEGF concentration at each time point divided by VEGF concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR versus PD).
Time Frame: Baseline to Day 1 of Weeks 3 through 53
Population: Safety population. Number of Participants analyzed = number of subjects with evaluable data and tumor response. n=number of subjects with evaluable data and tumor response at each specified time point. No subjects had PD following Week 33.
Measure: Median (Full Range); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 53
ratio
  Day 1, Week 3 (CR or PR, n=38) | 1.999 [0.42 to 19.96]
  Day 1, Week 3 (PD, n=15) | 1.948 [0.2 to 5.81]
  Day 1, Week 5 (CR or PR, n=37) | 1.383 [0.41 to 6.67]
  Day 1, Week 5 (PD, n=15) | 2.471 [0.09 to 10.93]
  Day 1, Week 7 (CR or PR, n=39) | 1.761 [0.4 to 8.56]
  Day 1, Week 7 (PD, n=13) | 1.405 [0.88 to 6.35]
  Day 1, Week 9 (CR or PR, n=37) | 2.215 [0.54 to 14.65]
  Day 1, Week 9 (PD, n=8) | 1.176 [0.32 to 5.6]
  Day 1, Week 13 (CR or PR, n=39) | 1.753 [0.33 to 21.39]
  Day 1, Week 13 (PD, n=2) | 3.921 [1.51 to 6.33]
  Day 1, Week 17 (CR or PR, n=36) | 2.012 [0.41 to 14.32]
  Day 1, Week 17 (PD, n=1) | 0.988 [0.988 to 0.988]
  Day 1, Week 21 (CR or PR, n=36) | 1.523 [0.24 to 8.75]
  Day 1, Week 21 (PD, n=1) | 1.510 [1.51 to 1.51]
  Day 1, Week 25 (CR or PR, n=35) | 1.809 [0.43 to 21.36]
  Day 1, Week 25 (PD, n=1) | 1.433 [1.433 to 1.433]
  Day 1, Week 29 (CR or PR, n=30) | 1.805 [0.4 to 6.04]
  Day 1, Week 29 (PD, n=1) | 1.929 [1.929 to 1.929]
  Day 1, Week 33 (CR or PR, n=31) | 2.248 [0.4 to 6.86]
  Day 1, Week 33 (PD, n=1) | 1.063 [1.063 to 1.063]
  Day 1, Week 37 (CR or PR, n=28) | 2.179 [0.59 to 7.15]
  Day 1, Week 41 (CR or PR, n=28) | 1.864 [0.51 to 7.84]
  Day 1, Week 45 (CR or PR, n=27) | 2.240 [0.22 to 8.81]
  Day 1, Week 49 (CR or PR, n=24) | 2.707 [0.75 to 8.24]
  Day 1, Week 53 (CR or PR, n=19) | 2.863 [0.66 to 15.81]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 3 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8519, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 5 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5879, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 7 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4757, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 9 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.1933, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 13 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4187, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 17 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3795, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 21 (CR or PR Versus PD); Test type: Superiority or Other; p = 1.0000, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 25 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.6333, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 29 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8679, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 33 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5920, Wilcoxon Rank Sum Test

21. Secondary Outcome: VEGF Ratio to Baseline Stratified by Tumor Response (CR or PR or [SD > = 12 Weeks] Versus PD)
Description: Median VEGF concentration at each time point divided by VEGF concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR or [SD > = 12 weeks] versus PD).
Time Frame: Baseline to Day 1 of Weeks 3 through 53
Population: as for outcome 20
Measure: Median (Full Range); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 98
ratio
  Day 1, Week 3 (CR or PR or SD, n=83) | 2.127 [0.3 to 19.96]
  Day 1, Week 3 (PD, n=15) | 1.948 [0.2 to 5.81]
  Day 1, Week 5 (CR or PR or SD, n=81) | 1.574 [0.24 to 24.75]
  Day 1, Week 5 (PD, n=15) | 2.471 [0.09 to 10.93]
  Day 1, Week 7 (CR or PR or SD, n=84) | 1.798 [0.3 to 10.01]
  Day 1, Week 7 (PD, n=13) | 1.405 [0.88 to 6.35]
  Day 1, Week 9 (CR or PR or SD, n=83) | 2.481 [0.35 to 17.14]
  Day 1, Week 9 (PD, n=8) | 1.176 [0.32 to 5.6]
  Day 1, Week 13 (CR or PR or SD, n=85) | 1.890 [0.28 to 21.39]
  Day 1, Week 13 (PD, n=2) | 3.921 [1.51 to 6.33]
  Day 1, Week 17 (CR or PR or SD, n=76) | 2.070 [0.26 to 14.23]
  Day 1, Week 17 (PD, n=1) | 0.988 [0.988 to 0.988]
  Day 1, Week 21 (CR or PR or SD, n=68) | 1.972 [0.24 to 10.66]
  Day 1, Week 21 (PD, n=1) | 1.510 [1.51 to 1.51]
  Day 1, Week 25 (CR or PR or SD, n=65) | 1.906 [0.43 to 21.36]
  Day 1, Week 25 (PD, n=1) | 1.433 [1.433 to 1.433]
  Day 1, Week 29 (CR or PR or SD, n=53) | 1.831 [0.4 to 8.18]
  Day 1, Week 29 (PD, n=1) | 1.929 [1.929 to 1.929]
  Day 1, Week 33 (CR or PR or SD, n=53) | 2.200 [0.4 to 6.86]
  Day 1, Week 33 (PD, n=1) | 1.063 [1.063 to 1.063]
  Day 1, Week 37 (CR or PR or SD, n=48) | 2.201 [0.53 to 8.76]
  Day 1, Week 41 (CR or PR or SD, n=48) | 1.859 [0.51 to 144.13]
  Day 1, Week 45 (CR or PR or SD, n=41) | 2.484 [0.22 to 8.81]
  Day 1, Week 49 (CR or PR or SD, n=37) | 2.329 [0.75 to 8.24]
  Day 1, Week 53 (CR or PR or SD, n=29) | 2.431 [0.66 to 15.81]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 3 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.6939, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 5 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.5871, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 7 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.4572, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 9 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.1120, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 13 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.4896, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 17 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.2369, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 21 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.6709, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 25 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.6382, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 29 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.8481, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 33 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3731, Wilcoxon Rank Sum Test

22. Secondary Outcome: Soluble VEGF Receptor 2 (sVEGFR2) Concentration at Baseline
Time Frame: Baseline
Population: Safety population. Number of Participants analyzed = number of subjects with evaluable data at baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 113
pg/mL | 9163.4 (2215.8)

23. Secondary Outcome: sVEGFR2 at Baseline Stratified by Tumor Response (CR or PR Versus PD)
Description: Summary statistics of sVEGFR2 at baseline by group (CR or PR versus PD) are presented.
Time Frame: Baseline (Cycle 1, Day 1)
Population: Safety population. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 56
pg/mL
  Cycle 1, Day 1 (CR or PR, n=40) | 9968.000 [3612 to 14080]
  Cycle 1, Day 1 (PD, n=16) | 8342.750 [5838.5 to 13987.5]
Statistical Analysis 1: Comparison: Sunitinib; CR or PR Versus PD; Test type: Superiority or Other; p = 0.0292, Wilcoxon Rank Sum Test

24. Secondary Outcome: sVEGFR2 at Baseline Stratified by Tumor Response (CR or PR or [SD > = 12 Weeks] Versus PD)
Description: Summary statistics of sVEGFR2 at baseline by group (CR or PR or SD versus PD) are presented.
Time Frame: Baseline (Cycle 1, Day 1)
Population: Safety population. n=number of subjects with levels of soluble protein biomarkers and tumor response at baseline.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 101
pg/mL
  Cycle 1, Day 1 (CR or PR or SD, n=85) | 9772.500 [3612 to 14080]
  Cycle 1, Day 1 (PD, n=16) | 8342.750 [5838.5 to 13987.5]
Statistical Analysis 1: Comparison: Sunitinib; CR or PR or (SD > = 12 Weeks) Versus PD; Test type: Superiority or Other; p = 0.1087, Wilcoxon Rank Sum Test

25. Secondary Outcome: sVEGFR2 Ratio to Baseline at Each Time Point
Description: sVEGFR2 concentration at each time point divided by sVEGFR2 concentration at baseline (ratio to baseline).
Time Frame: Baseline to Day 1 of Weeks 3 through 53
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 113
ratio
  Day 1, Week 3 (n=106) | 0.7 (0.2)
  Day 1, Week 5 (n=104) | 0.6 (0.2)
  Day 1, Week 7 (n=101) | 0.6 (0.2)
  Day 1, Week 9 (n=95) | 0.6 (0.2)
  Day 1, Week 13 (n=91) | 0.6 (0.2)
  Day 1, Week 17 (n=79) | 0.6 (0.2)
  Day 1, Week 21 (n=69) | 0.6 (0.2)
  Day 1, Week 25 (n=68) | 0.6 (0.2)
  Day 1, Week 29 (n=55) | 0.6 (0.2)
  Day 1, Week 33 (n=55) | 0.6 (0.2)
  Day 1, Week 37 (n=50) | 0.6 (0.2)
  Day 1, Week 41 (n=48) | 0.6 (0.2)
  Day 1, Week 45 (n=42) | 0.6 (0.2)
  Day 1, Week 49 (n=38) | 0.6 (0.2)
  Day 1, Week 53 (n=31) | 0.7 (0.2)

26. Secondary Outcome: sVEGFR2 Ratio to Baseline Stratified by Tumor Response (CR or PR Versus PD)
Description: Median sVEGFR2 concentration at each time point divided by sVEGFR2 concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR versus PD).
Time Frame: Baseline to Day 1 of Weeks 3 through 53
Population: as for outcome 20
Measure: Median (Full Range); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 40
ratio
  Day 1, Week 3 (CR or PR, n=39) | 0.704 [0.54 to 1.19]
  Day 1, Week 3 (PD, n=15) | 0.653 [0.52 to 1.37]
  Day 1, Week 5 (CR or PR, n=38) | 0.638 [0.36 to 0.97]
  Day 1, Week 5 (PD, n=15) | 0.531 [0.37 to 0.89]
  Day 1, Week 7 (CR or PR, n=40) | 0.596 [0.32 to 1.04]
  Day 1, Week 7 (PD, n=13) | 0.574 [0.38 to 0.9]
  Day 1, Week 9 (CR or PR, n=38) | 0.562 [0.28 to 1.34]
  Day 1, Week 9 (PD, n=8) | 0.603 [0.39 to 1.48]
  Day 1, Week 13 (CR or PR, n=40) | 0.555 [0.18 to 0.89]
  Day 1, Week 13 (PD, n=2) | 0.529 [0.51 to 0.55]
  Day 1, Week 17 (CR or PR, n=37) | 0.545 [0.23 to 0.93]
  Day 1, Week 17 (PD, n=1) | 0.687 [0.687 to 0.687]
  Day 1, Week 21 (CR or PR, n=36) | 0.566 [0.31 to 0.93]
  Day 1, Week 21 (PD, n=1) | 0.540 [0.54 to 0.54]
  Day 1, Week 25 (CR or PR, n=36) | 0.564 [0.29 to 0.96]
  Day 1, Week 25 (PD, n=1) | 0.509 [0.509 to 0.509]
  Day 1, Week 29 (CR or PR, n=30) | 0.564 [0.28 to 0.86]
  Day 1, Week 29 (PD, n=1) | 0.671 [0.671 to 0.671]
  Day 1, Week 33 (CR or PR, n=32) | 0.547 [0.24 to 0.91]
  Day 1, Week 33 (PD, n=1) | 0.610 [0.61 to 0.61]
  Day 1, Week 37 (CR or PR, n=29) | 0.554 [0.39 to 0.96]
  Day 1, Week 41 (CR or PR, n=29) | 0.561 [0.39 to 0.93]
  Day 1, Week 45 (CR or PR, n=28) | 0.535 [0.34 to 1.05]
  Day 1, Week 49 (CR or PR, n=25) | 0.555 [0.35 to 0.9]
  Day 1, Week 53 (CR or PR, n=20) | 0.630 [0.36 to 0.85]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 3 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3386, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 5 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.1949, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 7 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.7037, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 9 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5748, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 13 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.7470, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 17 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.4703, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 21 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.8162, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 25 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.5465, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 29 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.3495, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 33 (CR or PR Versus PD); Test type: Superiority or Other; p = 0.6397, Wilcoxon Rank Sum Test

27. Secondary Outcome: sVEGFR2 Ratio to Baseline Stratified by Tumor Response (CR or PR or [SD > = 12 Weeks] Versus PD)
Description: Median sVEGFR2 concentration at each time point divided by sVEGFR2 concentration at baseline (ratio to baseline) for subjects with tumor response (CR or PR or [SD > = 12 weeks] versus PD).
Time Frame: Baseline to Day 1 of Weeks 3 through 53
Population: as for outcome 20
Measure: Median (Full Range); unit: ratio
Arm/Group | Sunitinib
Number analyzed (Participants) | 96
ratio
  Day 1, Week 3 (CR or PR or SD, n=81) | 0.691 [0.29 to 1.54]
  Day 1, Week 3 (PD, n=15) | 0.653 [0.52 to 1.37]
  Day 1, Week 5 (CR or PR or SD, n=81) | 0.625 [0.31 to 1.36]
  Day 1, Week 5 (PD, n=15) | 0.531 [0.37 to 0.89]
  Day 1, Week 7 (CR or PR or SD, n=84) | 0.599 [0.31 to 1.3]
  Day 1, Week 7 (PD, n=13) | 0.574 [0.38 to 0.9]
  Day 1, Week 9 (CR or PR or SD, n=83) | 0.563 [0.15 to 1.34]
  Day 1, Week 9 (PD, n=8) | 0.603 [0.39 to 1.48]
  Day 1, Week 13 (CR or PR or SD, n=85) | 0.534 [0.18 to 1.4]
  Day 1, Week 13 (PD, n=2) | 0.529 [0.51 to 0.55]
  Day 1, Week 17 (CR or PR or SD, n=77) | 0.524 [0.23 to 1.25]
  Day 1, Week 17 (PD, n=1) | 0.687 [0.687 to 0.687]
  Day 1, Week 21 (CR or PR or SD, n=67) | 0.548 [0.26 to 1.39]
  Day 1, Week 21 (PD, n=1) | 0.540 [0.54 to 0.54]
  Day 1, Week 25 (CR or PR or SD, n=66) | 0.570 [0.29 to 1.28]
  Day 1, Week 25 (PD, n=1) | 0.509 [0.509 to 0.509]
  Day 1, Week 29 (CR or PR or SD, n=53) | 0.556 [0.28 to 1.19]
  Day 1, Week 29 (PD, n=1) | 0.671 [0.671 to 0.671]
  Day 1, Week 33 (CR or PR or SD, n=54) | 0.569 [0.24 to 1.24]
  Day 1, Week 33 (PD, n=1) | 0.610 [0.61 to 0.61]
  Day 1, Week 37 (CR or PR or SD, n=49) | 0.559 [0.31 to 1.54]
  Day 1, Week 41 (CR or PR or SD, n=48) | 0.572 [0.29 to 1.17]
  Day 1, Week 45 (CR or PR or SD, n=42) | 0.538 [0.34 to 1.2]
  Day 1, Week 49 (CR or PR or SD, n=38) | 0.569 [0.33 to 1.76]
  Day 1, Week 53 (CR or PR or SD, n=30) | 0.638 [0.36 to 1.56]
Statistical Analysis 1: Comparison: Sunitinib; Day 1, Week 3 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.4632, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib; Day 1, Week 5 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.1701, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Sunitinib; Day 1, Week 7 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.8204, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Sunitinib; Day 1, Week 9 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.5162, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: Sunitinib; Day 1, Week 13 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.9437, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: Sunitinib; Day 1, Week 17 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.4013, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: Sunitinib; Day 1, Week 21 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.9595, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: Sunitinib; Day 1, Week 25 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.6249, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: Sunitinib; Day 1, Week 29 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.3731, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: Sunitinib; Day 1, Week 33 (CR or PR or [SD > = 12 Weeks] Versus PD); Test type: Superiority or Other; p = 0.8263, Wilcoxon Rank Sum Test

28. Secondary Outcome: Patient-Assessed Fatigue
Description: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Scale: Overall score from 13-question questionnaire (measures fatigue/asthenia for patients with chronic, life-threatening illnesses). For each question, patient rates condition for the past week on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Total FACIT-Fatigue score = sum score of the 13 question scores; total range: 0 - 52; higher total score represents less fatigue. End of treatment assessment was for subjects who completed the study only.
Time Frame: Baseline (Day 1, Week 1), Day 1 of Weeks 3, 5, 7, 9, 11, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, Week 53 (End of Treatment)
Population: Safety population. Number of Participants analyzed = number of subjects evaluable for the FACIT-Fatigue analysis. n=number of subjects with scores at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 118
scores on a scale
  Baseline (n=118) | 39.29 (9.55)
  Week 3 (n=113) | 36.98 (11.38)
  Week 5 (n=110) | 35.44 (10.87)
  Week 7 (n=106) | 36.54 (10.86)
  Week 9 (n=97) | 36.82 (9.43)
  Week 11 (n=93) | 35.94 (9.75)
  Week 13 (n=90) | 36.58 (10.32)
  Week 17 (n=80) | 37.44 (9.83)
  Week 21 (n=71) | 38.42 (10.08)
  Week 25 (n=62) | 38.05 (9.69)
  Week 29 (n=60) | 36.77 (10.89)
  Week 33 (n=55) | 36.00 (11.22)
  Week 37 (n=52) | 37.88 (9.77)
  Week 41 (n=50) | 36.96 (10.74)
  Week 45 (n=42) | 38.71 (8.66)
  Week 49 (n=41) | 39.32 (8.98)
  Week 53 (End of Treatment) (n=40) | 39.05 (8.62)

29. Secondary Outcome: Cancer Related Symptoms, Well-Being, and Concerns
Description: FACT-Advanced Kidney Cancer Symptom Index (FKSI) Questionnaire: subscale designed to be a stand-alone instrument to measure symptoms and quality of life in patients with advanced kidney cancer. Contains 15 questions. Each question was answered on a 5-point Likert-type scale ranging from 0 to 4 (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). Total FKSI score = sum score of the 15 item scores; total range: 0 - 60; 0 (most severe symptoms and concerns) to 60 (no symptoms or concerns). End of treatment assessment was for subjects who completed the study only.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 109
scores on a scale
  Baseline (n=109) | 44.68 (7.78)
  Week 3 (n=104) | 43.69 (8.38)
  Week 5 (n=101) | 42.71 (8.64)
  Week 7 (n=97) | 43.69 (7.99)
  Week 9 (n=88) | 44.11 (7.55)
  Week 11 (n=84) | 43.26 (7.88)
  Week 13 (n=81) | 43.49 (8.01)
  Week 17 (n=72) | 44.21 (7.34)
  Week 21 (n=63) | 45.51 (7.50)
  Week 25 (n=55) | 45.42 (8.00)
  Week 29 (n=55) | 44.64 (8.42)
  Week 33 (n=50) | 44.06 (8.35)
  Week 37 (n=47) | 45.23 (8.03)
  Week 41 (n=45) | 44.71 (8.16)
  Week 45 (n=37) | 46.73 (6.94)
  Week 49 (n=36) | 45.92 (7.31)
  Week 53 (End of Treatment) (n=35) | 45.94 (7.29)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 45/119
Other Adverse Events (participants affected / at risk) | 117/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=119)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Large intestinal obstruction (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Catheter related complication (General disorders) | 1
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Disease progression (General disorders) | 8
Gait disturbance (General disorders) | 1
Oedema (General disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Eastern cooperative oncology group performance status worsened (Investigations) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=119)
Anaemia (Blood and lymphatic system disorders) | 26
Neutropenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Hypothyroidism (Endocrine disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 18
Abdominal pain upper (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 62
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 18
Gastritis (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6
Gingivitis (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 35
Stomatitis (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 26
Asthenia (General disorders) | 26
Face oedema (General disorders) | 12
Fatigue (General disorders) | 42
Mucosal inflammation (General disorders) | 37
Oedema (General disorders) | 9
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 10
Blood alkaline phosphatase increased (Investigations) | 7
Blood creatinine increased (Investigations) | 13
Lipase increased (Investigations) | 10
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 18
Weight decreased (Investigations) | 18
White blood cell count decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 32
Headache (Nervous system disorders) | 13
Neuropathy peripheral (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Hair colour changes (Skin and subcutaneous tissue disorders) | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 49
Periorbital oedema (Skin and subcutaneous tissue disorders) | 8
Petechiae (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 20
Skin discolouration (Skin and subcutaneous tissue disorders) | 27
Yellow skin (Skin and subcutaneous tissue disorders) | 15
Hypertension (Vascular disorders) | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.